CLINICAL TRIAL: NCT05179525
Title: An Open-Label, One-Sequence Study to Evaluate the Steady- State Comparative Bioavailability of Intramuscular Risperidone ISM® and EU Risperdal® (Sourced From Germany)
Brief Title: Comparative Bioavailability of Risperidone.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rovi Pharmaceuticals Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ROV-RISP-2020-01
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Schizophrenia
Keywords: risperidone; schizophrenia; long-acting injectable
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; Tablets

STUDY DESIGN:
Intervention Model Description: This is an open-label, 1-sequence study to Evaluate the Steady- State Comparative Bioavailability of Intramuscular Risperidone ISM® and EU Risperdal® (Sourced From Germany) in subjects with schizophrenia who are on stable oral risperidone treatment. The study consists of a screening visit, 1 treatment period with inpatient and outpatient visits, and a follow-up visit.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Risperidone ISM® 100 mg (Experimental): Subjects will receive 4 mg oral risperidone once daily for 7 days. After the 1 week oral risperidone regimen subjects will be administered 100 mg risperidone ISM as an injectable into the gluteal muscle. A total of 4 doses of intramuscular (IM) 100 mg risperidone ISM® will be administered deeply into the gluteal muscle. Each dose will be separated by 4 weeks.
  Interventions: Drug: Risperidone ISM® 100 mg; Drug: Risperdal 4mg Tablet

INTERVENTIONS:
Drug: Risperidone ISM® 100 mg — 100 mg of risperidone ISM® administered every 4 weeks
Drug: Risperdal 4mg Tablet — 4 mg oral risperidone once daily for 7 days

SUMMARY:
This is an Open-Label, One-Sequence Study to Evaluate the Steady- State Comparative Bioavailability of Intramuscular Risperidone ISM® and EU Risperdal® (Sourced From Germany).

DETAILED DESCRIPTION:
This was an open-label, 1-sequence study in patients who are were stable oral risperidone treatment. The study consisted of a screening visit, 1 treatment period with inpatient and outpatient visits, and a Follow-up visit.

Patients who were receiving existing oral risperidone treatment (4 mg) continued the oral regimen for 1 week to achieve steady-state concentrations of risperidone (Treatment A). Following the oral risperidone treatment, a single IM dose of 100 mg Risperidone ISM® was administered deeply into the gluteal muscle. A total of 4 IM doses were given, each dose separated by 4 weeks (Treatment B).

Safety assessments and PK sampling were performed once each dosing day and each outpatient visit. A final Follow-up visit was conducted to assess each patient for safety and to obtain PK samples.

Approximately 80 (with no screening failure) patients were planned for enrolment, with the intent to complete 48 patients with the assumption of an approximate drop-out/not valuable PK rate of 40%.

The primary objective of this study was to evaluate the steady-state comparative bioavailability of 100 mg Risperidone ISM® injectable every 4 weeks compared to once-daily 4 mg oral risperidone in patients with schizophrenia stabilized on oral risperidone treatment.

The secondary objective of this study was to evaluate the safety and tolerability of 100 mg Risperidone ISM® injectable every 4 weeks compared to once-daily 4 mg oral risperidone in patients with schizophrenia stabilized on oral risperidone treatment.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be considered eligible to participate in this study if each one of the following inclusion criteria is satisfied at screening (or at baseline when specified):

1. Male or female aged ≥18 and <65 years with a body mass index (BMI) of ≥17 kg/m2 but ≤35 kg/m2
2. Current diagnosis of schizophrenia, according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria
3. Outpatient; not hospitalized for worsening of schizophrenia within the last 3 months (hospitalization for social management within this time period is acceptable)
4. Medically stable over the last month and psychiatrically stable without significant symptom exacerbation over the last 3 months based on the investigator's judgement
5. On oral risperidone 4 mg daily as maintenance therapy for at least the last 4 weeks prior to screening and on 4 mg oral risperidone once daily QD for at least one week prior baseline (Day1, Visit 2)
6. Agrees to taper off all prohibited medications prior to baseline
7. On a stable dosage of all permitted medications (with the exception of medication to be used on an as-needed basis) for at least 2 weeks prior to the baseline visit and for the duration of the study
8. Clinical Global Impression - Severity (CGI-S) score of ≤4 (moderately ill)
9. A female subject of childbearing potential who is sexually active and using a medically accepted contraceptive method. Acceptable methods include condoms (male or female) with or without spermicidal agent, diaphragm or cervical cap with spermicide, medically prescribed intrauterine device, and hormonal contraceptives. A female subject of childbearing potential who is not currently sexually active must agree that should she be so while participating in the trial, she will use a medically accepted method of contraception for the remainder of the study and for 1 month afterward. Female patients who have had a hysterectomy, bilateral tubal ligation, or bilateral salpingooophorectomy are considered surgically sterile and are thus are exempt from the requirement to use contraception. Female patients who are postmenopausal are considered not of childbearing potential and thus exempt from the contraception requirement; for the purpose of this study, postmenopausal is defined as the permanent cessation of menstruation for at least 12 months prior to screening in women ≥ 45 years of age.
10. Female subjects must have a negative pregnancy test at screening (serum test) and baseline (urine test)
11. Psychotherapy should not be started or changed during a patient's participation in the study. It is acceptable for a patient already receiving psychotherapy to participate in the study
12. Able to speak, read, and understand sufficiently to allow completion of all study assessments
13. Must provide written informed consent prior to the initiation of any protocol-specific procedures

Exclusion Criteria:

Subjects will not be considered eligible to participate in this study if any one of the following exclusion criteria is satisfied at screening (or at baseline when specified):

1. Presence of an uncontrolled, unstable, clinically significant medical condition (eg, renal, endocrine, hepatic, respiratory, cardiovascular, hematologic, immunologic or cerebrovascular disease, or malignancy) that in the opinion of the investigator could have interfered with the interpretation of safety and PK evaluations
2. Presence of a clinically significant vital sign or physical examination finding that in the opinion of the investigator could potentially interfere with the ability to evaluate safety and tolerability of the trial medication or could impair the subject's ability to complete the trial
3. Presence of a clinically significant abnormality on blood or urine safety tests, which do not improve on retesting. In particular, laboratory and/or clinical evidence of clinically significant hepatic conditions, such as:

   * alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 × upper limit of normal (ULN) and total bilirubin > 2 × ULN; or
   * ALT or AST > 3 × ULN with the appearance of jaundice, worsening of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, or eosinophilia
4. Corrected QT interval, Fridericia's correction (QTcF) interval greater than 450 msec for males and 470 msec for females, or other clinically significant ECG abnormality on screening or baseline
5. If female, a positive serum pregnancy test, or planning to become pregnant between signing informed consent and 1 month after the last dose of trial medication, or is breastfeeding a child
6. Uncontrolled or unstable diabetes, or a clinically significant abnormal Hba1c blood level
7. Known or suspected (non-febrile) seizure disorder
8. Known serological evidence of human immunodeficiency (HIV) antibody
9. History of hepatitis B infection within the past year, or history of hepatitis C infection that has not been adequately treated and abnormal LFT values.
10. History of neuroleptic malignant syndrome
11. Current or past history of clinically significant tardive dyskinesia
12. Primary diagnosis other than schizophrenia diagnosis that is primarily responsible for current symptoms and functional impairment
13. Known or suspected diagnosis of mental retardation or organic brain disorder
14. Positive urine drug/alcohol (ethanol breathalyzer is also acceptable) screen finding, unless the positive finding can be accounted for by documented prescription use.

    Individuals who have positive results for alcohol, cannabis, or other psychotropic substances but are not dependent on or abusing these substances may be included at the investigator's discretion, following a discussion between the investigator and the medical monitor
15. Heavy smoker (consumption of >40 cigarettes daily)
16. Fulfillment of the DSM-5 criteria for moderate or severe substance use disorder (excluding nicotine) within the past 6 months
17. Diagnosis of a psychotic disorder or a behavioral disturbance that is thought to be substance-induced or due to substance abuse
18. In the investigator's opinion, at imminent risk of committing self-harm or harm to others, based on clinical interview and responses provided on the C-SSRS. Individuals will be excluded if they report having suicidal ideation of Type 4 or 5 in the past 2 months, or suicidal behavior in the past 6 months, as measured by the C-SSRS at screening or baseline
19. On more than 1 antidepressant; or if on just one, a change in dose within the last 4 weeks prior to screen
20. Use of depot antipsychotics within the last 6 to 9 months
21. Use of electroconvulsive therapy (ECT) within the last 3 months
22. Use of moderate or strong cytochrome P450 (CYP) 3A4 enzyme inducers and inhibitors (carbamazepine, phenytoin, rifampicin, phenobarbital) or moderate or strong CYP2D6 inhibitors (fluoxetine, paroxetine) (see Appendix 11.2) within 3 days or a time period of 5 half lives of the concerning drug, whichever is longer, prior to baseline
23. Unwilling to discontinue any of prohibited medications prior to the baseline visit; or, in the opinion of the investigator, is unable to safely taper off such medication without significant destabilization or increased risk of self-harm (suicide). Prohibited medications may include antipsychotics, phenobarbital, fluoxetine, fluoxetine combinations, paroxetine, benzodiazepines except lorazepam, diazepam, oxazepam, psychotropics, herbal drugs/dietary supplements for depression, anxiety, insomnia, rifampicin, and quinidine
24. Receipt of any investigational drugs within the last 3 months
25. Current participation in any other clinical trial
26. In the investigator's opinion, medically non-compliant in the management of his or her disease
27. Known or suspected allergy or hypersensitivity to risperidone or any of the ISM excipients
28. Previous non-responder to risperidone treatment
29. Currently under involuntary in-patient commitment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2021-09-17 (Actual)

PRIMARY OUTCOMES:
Area under the curve during the dosing interval (AUCtau) | 28-day period following administration of the fourth dose of risperidone ISM®
  Mean steady-state area under the curve during the dosing interval for the active moiety

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Llaudó, MD, Study Chair — Laboratorios Farmacéuticos Rovi
Locations (4):
- United States (4):
  - Collaborative NeuroScience Research, LLC, Garden Grove, California
  - CBH Health, LLC, Gaithersburg, Maryland
  - Hassman Research Institute, Berlin, New Jersey
  - Rajinder Shiwach, DeSoto, Texas

IPD SHARING:
Plan to Share IPD: No